CLINICAL TRIAL: NCT05088668
Title: The Effectiveness of Augmented Reality Combined With Scapular Repositioning Exercises in Patients With Chronic Shoulder Pain and Scapular Dyskinesis: a Randomized Clinical Trial
Brief Title: Augmented Reality for Shoulder Pain and Scapular Dyskinesis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistic issues
Sponsor: Ruben Fernandez Matias (Other)
Responsible Party: Sponsor-Investigator, Ruben Fernandez Matias, Clinical Professor, University of Alcala
Organization: University of Alcala (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25072021
Record Dates: First submitted 2021-09-19; First posted 2021-10-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The researchers involved in measuring outcomes will not be aware of treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Agumented Reality combined with scapular exercises (Experimental): Scapular exercises performed with glasses of augmented reality during sessions at clinic, and without glasses at home.
  Interventions: Other: Augmented reality; Other: Scapular repositioning exercise
- Scapular exercises (Active Comparator): Scapular exercises performed all the time without glasses.
  Interventions: Other: Scapular repositioning exercise

INTERVENTIONS:
Other: Augmented reality — The subjects will perform scapular repositioning exercise using glasses of augmented reality to see their scapular movement simultaneously. Furthermore, they will also see at the same time a video record of an "ideal" scapular movement, and will me encouraged to simulate that "ideal" scapular movement.
  Arms: Agumented Reality combined with scapular exercises
Other: Scapular repositioning exercise — Subjects will perform scapular repositioning exercises for improving scapular movement.

SUMMARY:
The aim of this study is to analyze whether an Augmented Reality based scapular stabilization exercise program is more effective than conventional programs in patients with chronic shoulder pain and Scapular Dyskinesis.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral mechanical shoulder pain of nonspecific origin (non-traumatic) lasting at least 3 months.
* Weakness in flexion, abduction and/or external rotation isometric strength testing.
* Presence of scapular dyskinesis according to Kibler, Scapular Assistance Test, and Scapular Reposition Test.

Exclusion Criteria:

* Previous shoulder surgery.
* History of shoulder fracture or glenohumeral luxation.
* History of acromioclavicular joint injury.
* Presence of massive rotator cuff rears.
* Presence of frozen shoulder.
* Cervical hernias or radiculopathy.
* Fibromyalgia.
* Neuropathic pain.
* Cervical and/or vestibular problems with dizziness, unsteadiness, or vertigo.
* Medical contraindication for performing exercise (cardio-vascular or cardio-pulmonar diseases, systemic diseases, metabolic diseases in non-controlled acute state).
* Blindness.
* Actually being treated with physical therapy for shoulder pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Pain intensity measured with a visual analogue scale which ranges from 0 (no pain) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Change in shoulder disability | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Shoulder disability measured with Shoulder Pain and Disability Index (SPADI), which ranges from 0 (no disability) to 100 (maximum degree of disability).
Change in arm disability | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Arm disability measured with Disabilities of the Arm, Shoulder, and Hand (Quick-DASH), which ranges from 0 (no disability) to 100 (maximum degree of disability).
Change in kinesiophobia | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Kinesiophobia measured with Tampa Scale of Kinesiophobia (TSK-11), which ranges from 0 (no kinesiophobia) to 100 (maximum degree of kinesiophobia)
Change in catastrophism | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Pain catastrophism measured with Pain Catastrophism Scale (PCS), which ranges from 0 (no catastrophism) to 100 (severe catastrophism).
Change in shoulder range of motion | Baseline, 1-month, 2-months, 3-months, and 6-months
  Shoulder range of motion in abduction, flexion, internal and external rotation, measured with a goniometer
Change in surface electromiography | Baseline, change from baseline at 1-month, change from baseline at 2-months, change from baseline at 3-months, and change from baseline at 6-months
  Electromiographic activity of serratus anterior, upper trapezius, lower trapezius, and deltoid medimum muscles. Percent of electromiographic activity as a function of maximum voluntary isometric contraction, as well as latency of muscle activation during scaption will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruben Fernandez-Matias, Alcalá de Henares, Spain